CLINICAL TRIAL: NCT01815879
Title: Metastatic Colorectal Cancer Liver Metastases Outcomes After Resin 90Y Microsphere Radioembolization in the USA Evaluation Project
Acronym: MORE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Andrew Kennedy (Industry)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor-Investigator, Andrew Kennedy, Principal Investigator and Sponsor-Investigator, Sarah Cannon
Organization: Sarah Cannon (Industry)
Other Study IDs: MORE
Record Dates: First submitted 2012-12-18; First posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: metastatic colorectal cancer; liver metastases; 90Y resin microsphere radioembolization; retrospective data analysis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Control Group: Retrospective review of clinical data on at least 1,000 evaluable US patients with 12+weeks follow up that were treated with 90Y resin microsphere radioembolization for metastatic colorectal liver metastases

SUMMARY:
Investigator initiated multi-institutional retrospective review of clinical and radiographic outcomes after 90Y resin microsphere radioembolization for metastatic colorectal liver metastases in the USA. The target is for at least 1,000 evaluable patients with 12+ weeks follow up.

DETAILED DESCRIPTION:
Investigator initiated multi-institutional retrospective review of clinical and radiographic outcomes after 90Y resin microsphere radioembolization for metastatic colorectal liver metastases in the USA. The target is for at least 1,000 evaluable patients with 12+ weeks follow up. Objectives:

Independent data collection and reporting of pre treatment and 12 week post treatment clinical, radiographic and radiation parameters and outcomes in patients treated in the USA from 2002-2010. Data beyond 12 weeks will be collected and highly desirable, however as a minimum all patients will have 12 week follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received 90Y resin microsphere radioembolization for metastatic colorectal cancer with liver metastases between November 2010 and March 2011 in the USA. Patients must have at least 12 weeks of follow up.

Exclusion Criteria:

* Patients who received glass 90Y microsphere radioembolization for metastatic colorectal liver metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal liver metastases in the USA treated with 90Y resin microsphere radioembolization
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events at day 0-90 post 90Y therapy using CTCae 3.0 criteria. | 3 months
  Multiple systems monitored for side effects possibly related to liver radiotherapy.

SECONDARY OUTCOMES:
Radiographic response rate at 90 days (+/- 45 days) from treatment day, compared to pretreatment scans. | 3 months
  Pretreatment planning scans (-45 to -1 day) compared to post radiotherapy scans of the liver, PET/CT not recommended, prefer MRI with Gd or CT with contrast, 3 phase, with rescanning in similar fashion at day 90 post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Kennedy, MD, FACRO, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Contact Sarah Cannon, Nashville, Tennessee, United States